CLINICAL TRIAL: NCT07281287
Title: Evaluating the Implementation and Impact of Standard-of-care Delivered Oncology Financial Navigation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Courtney Williams, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-300012763; 1K01CA296932 (NIH)
Record Dates: First submitted 2025-12-03; First posted 2025-12-15 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Oncology; Financial Toxicity; Counseling
Keywords: Financial Navigation; Out of pocket cost; Oncology; oncology Financial hardship
MeSH Terms: conditions — Neoplasms; Financial Stress

STUDY DESIGN:
Intervention Model Description: This will be a secondary data analysis of patient-reported data routinely collected since 2020 for patients with cancer seen at the UAB Medical Oncology clinic. All patients with data will be included in the analysis, as this is an evaluation of oncology financial navigation integration into real-world clinical teams. Therefore, due to a lack of comparable controls during the oncology financial navigation intervention, we will use historical controls matched by sociodemographic and cancer characteristics for comparison.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients receiving standard-of-care-delivered financial navigation (Experimental)
  Interventions: Behavioral: Financial navigation
- Historical control patients who did not receive financial navigation (No Intervention)

INTERVENTIONS:
Behavioral: Financial navigation — Oncology financial navigation is an evidence-based intervention which helps patients prepare for out-of-pocket treatment costs, optimize health insurance, and access financial resources to reduce cancer-related financial hardship.
  Arms: Patients receiving standard-of-care-delivered financial navigation

SUMMARY:
The purpose of this study is to understand the implementation and impact of a pragmatically-delivered oncology financial navigation program. The main questions it aims to answer are:

1. How did oncology financial navigation implementation strategies affect implementation outcomes?
2. What is the impact of financial navigation on patient financial hardship, quality of life, and psychological distress?
3. How were implementation strategies utilized to overcome barriers to oncology financial navigation?

Researchers will examine secondary, standard-of-care collected, patient-reported data, electronic medical record data, and qualitative interview data to answer these questions.

DETAILED DESCRIPTION:
Guided by the RE-AIM Extension for Equitable Sustainability framework, the investigators will use a series of implementation and effectiveness aims to evaluate equitable implementation of oncology financial navigation into routine cancer care delivery. The investigators hypothesize the proposed assessment will identify potential areas to improve implementation of oncology financial navigation, which will result in better financial and clinical outcomes for patients with cancer. The investigators propose a pragmatic, hybrid effectiveness-implementation study to assess outcomes of oncology financial navigation delivered as routine cancer care and collect information on strategies to address implementation barriers. Outcomes will be assessed overall and for inequities by race, residence, and insurance status using the following specific aims:

Aim 1. Track oncology financial navigation implementation strategies and their effect on implementation outcomes

Aim 2. Evaluate oncology financial navigation effectiveness

Aim 3. Assess how implementation strategies were utilized to overcome barriers to oncology financial navigation

ELIGIBILITY:
Aim 1:

Inclusion criteria: As oncology financial navigation will be implemented as standard of care, implementation outcomes will be evaluated for:

1. All patients with cancer seen at the University of Alabama at Birmingham (UAB) Medical Oncology clinic
2. UAB oncology financial navigators

Exclusion criteria: None.

Aim 2:

Inclusion criteria: This will be a secondary data analysis of patient-reported data routinely collected since 2020, which will include:

1. Patients with cancer seen at the UAB Medical Oncology clinic
2. Patients with non-missing patient-reported outcome data

Exclusion criteria: None.

Aim 3:

Inclusion criteria:

1. Patients who have received oncology financial navigation
2. Providers (oncology financial navigators, social workers, nurse managers, oncologists) involved with the oncology financial navigation program
3. Health system team members (billing specialists, cancer service line leadership) involved with the oncology financial navigation program

Exclusion criteria: None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in financial hardship | 6 months post-initiation of systemic therapy
  Change in patient-reported financial distress (COmprehensive Score for financial Toxicity)
Change in financial difficulties | 6 months post-initiation of systemic therapy
  Change in patient-reported financial difficulties (trouble paying for basic needs, utilities, transportation or lodging for treatment, medications, medical supplies, upfront medical payments, insurance or medical bills, child or eldercare, and employment or disability issues)
Change in quality of life | 6 months post-initiation of systemic therapy
  Change in patient-reported quality of life (PROMIS v1.1 Global Health)
Change in psychological distress | 6 months post-initiation of systemic therapy
  Change in patient-reported psychological distress (National Comprehensive Cancer Network Distress Thermometer)
Utilization of implementation strategies | Quarterly tracking of strategies with monthly assessment of implementation outcomes, through study completion, an average of 4 years
  Track oncology financial navigation implementation strategies using the Expert Recommendations for Implementing Change (ERIC) implementation strategy taxonomy and their effect on implementation outcomes of Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM)
Patient, provider, and health system perspectives of oncology financial navigation implementation barriers addressed via implementation strategies | Annually through study completion, an average of 4 years
  Using qualitative interviews, we will assess patient, provider, and health system perspectives of oncology financial navigation implementation barriers addressed via implementation strategies

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Williams, DrPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-02-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT07281287/Prot_SAP_ICF_000.pdf